CLINICAL TRIAL: NCT06372847
Title: Assessment of the Effect of Hypoglossal Nerve Stimulation Therapy on the Site of Collapse During DISE
Brief Title: DISE-HNS Effect Study
Acronym: DISE-HNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Project ID 6214
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Hypoglossal nerve stimulation; Drug-induced sleep endoscopy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Intervention Model Description: Before-and-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving hypoglossal nerve stimulation (HNS) (Other): All included patients will be part of this arm. Patients who are eligible for HNS-therapy for obstructive sleep apnea (OSA) will be invited to participate in the study. Data from the baseline PSG and baseline DISE as part of the standard pathway for HNS-eligibility will be accessed and collected. All patients will undergo HNS-implantation and receive HNS-therapy as part of the standard pathway. After one year of treatment, information from the one-year follow-up PSG as part of the standard pathway will be collected. Furthermore, patients will undergo an additional one-year follow-up DISE.
  Interventions: Device: Hypoglossal nerve stimulation implant; Diagnostic Test: Polysomnography; Procedure: Drug-induced sleep endoscopy (DISE)

INTERVENTIONS:
Device: Hypoglossal nerve stimulation implant — The hypoglossal nerve stimulation (HNS) implantation and therapy will be performed according to the standard clinical practice without additional procedures. Information about the surgical procedure will be collected. HNS implant information and settings will be collected throughout the study until the last study measurement (one year follow-up PSG and DISE) for that patient. No additional measures or interventions as part of the research project will be performed during implantation or treatment with HNS.
Diagnostic Test: Polysomnography — A PSG at one-year follow-up is part of the standard follow-up pathway in patients receiving HNS therapy. In this study, PSG data will be collected from both baseline and one-year follow-up PSGs to assess treatment effect. Additionally, PSG data will be used for non-invasive prediction of the site and pattern of collapse using a novel, validated tool developed at our research group.
Procedure: Drug-induced sleep endoscopy (DISE) — Drug-induced sleep endoscopy (DISE) is the clinical standard diagnostic test to assess site, pattern and degree of upper-airway collapse in OSA. Baseline DISE is part of the standard clinical pathway for HNS eligibility.
  In this study, DISE data will be collected from routine baseline DISE without any additional procedures for the patient. They will undergo an additional DISE at one-year follow-up to assess the effect of HNS-therapy on site, pattern and degree of collapse. Both DISEs will be performed according to routine clinical practice in the operating theatre. Sleep will be induced using 1.5 mg bolus injection midazolam and target-controlled propofol infusion (2.0 - 3.0 μg). A flexible fiberoptic nasopharyngoscope will be transnasally inserted. Site, pattern and degree of collapse will be assessed using a standardized scoring system. Other maneuvers, including chin-lift, the use of a simulation bite or lateral position of the head will be performed according to clinical practice.

SUMMARY:
The purpose of this study is to assess the site, pattern and degree of upper airway collapse before and during hypoglossal nerve stimulation (HNS) treatment using clinical standard drug-induced sleep endoscopy (DISE) and using a novel, non-invasive method predicting site of collapse from raw polysomnography (PSG) data.

Furthermore, outcomes will be compared between responders and non-responders.

DETAILED DESCRIPTION:
Patients who will receive hypoglossal nerve stimulation therapy will be recruited at the pre-operative consultation at the department of ENT. As part of the standard procedure, all patients who are eligible for HNS have already undergone DISE.

To be included in the study, the patient should have undergone or is scheduled to undergo a baseline PSG within two years of HNS implantation.

All patients will undergo HNS-implantation and receive HNS-therapy as part of the standard pathway.

One year after HNS-therapy, patients will undergo another PSG as part of routine practice in these patients. An additional DISE will be performed to assess the effect of HNS on the site, pattern and degree of upper airway collapse.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Eligible for HNS-therapy:
* AHI between 15 and 65 events/hour
* BMI under 32 kg/m2
* Absence of complete concentric collapse of palate (CCC) on DISE
* Intolerance or failure of continuous positive airway pressure (CPAP)-treatment
* Intolerance or failure of mandibular advancement device (MAD)-treatment
* Combination of central and mixed apneas less than 25% of total apneas on recent PSG (not older than two years)
* Scheduled for HNS-implantation at the Antwerp University Hospital
* Capable of giving informed consent
* Baseline polysomnography planned or performed in the last 2 years at the Antwerp University Hospital

Exclusion Criteria:

* Patients will not receive HNS-therapy at the Antwerp University Hospital
* Known medical history of intellectual disability, memory disorders or current psychiatric disorders (psychotic illness, major depression, or acute anxiety attacks as mentioned by the patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Δ%area-of-collapse at the level of the lateral walls | Between baseline and one year follow-up
  The percentage of the area of collapse at the level of the lateral walls - measured using DISE - will be calculated using ImageJ software. The percentage difference of collapse between baseline and one-year follow-up will be calculated.

SECONDARY OUTCOMES:
Δ%area-of-collapse at the level of the palate, tongue base and epiglottis | Between baseline and one year follow-up
  The percentage of the area of collapse at the level of the palate, tongue base and epiglottis - measured using DISE - will be calculated using ImageJ software. The percentage difference of collapse between baseline and one-year follow-up will be calculated.
Δ%area-of-collapse at each possible site of upper airway collapse (palate, lateral walls, tongue base, epiglottis) in responders and non-responders | Between baseline and one year follow-up
  The Δ%area-of-collapse will be specifically identified in the group of responders and the group of non-responders, to compare these two groups.
DISE-score during baseline DISE and during one-year follow-up DISE. | At baseline and at one-year follow-up
  DISE-scores (pattern and degree of collapse at each site of upper airway collapse) will be scored to assess the effect of HNS on this outcome.
Non-invasive site and pattern of collapse | At baseline and at one-year follow-up
  Non-invasive site and pattern of collapse assessed using the novel developed and validated tool at baseline and 1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier M Vanderveken, MD, PhD, Principal Investigator — Department of Otorhinolaryngology and Head & Neck Surgery, Antwerp University Hospital
Locations (1):
- Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No
All data will solely be available to members of the A-SLEAP research team (Antwerp University Hospital and University of Antwerp, led by the principal investigator of this study). Data will not be shared outside of the research team or the affiliated organizations.

REFERENCES:
- [Background] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535
- [Background] Somers VK, White DP, Amin R, Abraham WT, Costa F, Culebras A, Daniels S, Floras JS, Hunt CE, Olson LJ, Pickering TG, Russell R, Woo M, Young T; American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology; American Heart Association Stroke Council; American Heart Association Council on Cardiovascular Nursing; American College of Cardiology Foundation. Sleep apnea and cardiovascular disease: an American Heart Association/american College Of Cardiology Foundation Scientific Statement from the American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology, Stroke Council, and Council On Cardiovascular Nursing. In collaboration with the National Heart, Lung, and Blood Institute National Center on Sleep Disorders Research (National Institutes of Health). Circulation. 2008 Sep 2;118(10):1080-111. doi: 10.1161/CIRCULATIONAHA.107.189375. Epub 2008 Aug 25. No abstract available. PMID 18725495
- [Background] Marshall NS, Wong KK, Cullen SR, Knuiman MW, Grunstein RR. Sleep apnea and 20-year follow-up for all-cause mortality, stroke, and cancer incidence and mortality in the Busselton Health Study cohort. J Clin Sleep Med. 2014 Apr 15;10(4):355-62. doi: 10.5664/jcsm.3600. PMID 24733978
- [Background] Gottlieb DJ, Punjabi NM. Diagnosis and Management of Obstructive Sleep Apnea: A Review. JAMA. 2020 Apr 14;323(14):1389-1400. doi: 10.1001/jama.2020.3514. PMID 32286648
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Sullivan CE, Issa FG, Berthon-Jones M, Eves L. Reversal of obstructive sleep apnoea by continuous positive airway pressure applied through the nares. Lancet. 1981 Apr 18;1(8225):862-5. doi: 10.1016/s0140-6736(81)92140-1. PMID 6112294
- [Background] Vena D, Op de Beeck S, Mann D, et al. Pharyngeal site of collapse and collapsibility estimated from airflow predict oral appliance treatment efficacy. Sleep Medicine. 2022/12/01/ 2022;100:S264-S265. doi:https://doi.org/10.1016/j.sleep.2022.05.713
- [Background] Sutherland K, Vanderveken OM, Tsuda H, Marklund M, Gagnadoux F, Kushida CA, Cistulli PA. Oral appliance treatment for obstructive sleep apnea: an update. J Clin Sleep Med. 2014 Feb 15;10(2):215-27. doi: 10.5664/jcsm.3460. PMID 24533007
- [Background] Vanderveken OM, Beyers J, Op de Beeck S, Dieltjens M, Willemen M, Verbraecken JA, De Backer WA, Van de Heyning PH. Development of a Clinical Pathway and Technical Aspects of Upper Airway Stimulation Therapy for Obstructive Sleep Apnea. Front Neurosci. 2017 Sep 21;11:523. doi: 10.3389/fnins.2017.00523. eCollection 2017. PMID 28983236
- [Background] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- [Background] Vanderveken OM, Maurer JT, Hohenhorst W, Hamans E, Lin HS, Vroegop AV, Anders C, de Vries N, Van de Heyning PH. Evaluation of drug-induced sleep endoscopy as a patient selection tool for implanted upper airway stimulation for obstructive sleep apnea. J Clin Sleep Med. 2013 May 15;9(5):433-8. doi: 10.5664/jcsm.2658. PMID 23674933
- [Background] Huyett P, Kent DT, D'Agostino MA, Green KK, Soose RJ, Kaffenberger TM, Woodson BT, Huntley C, Boon MS, Heiser C, Birk A, Suurna MV, Lin HS, Waxman JA, Kezirian EJ. Drug-Induced Sleep Endoscopy and Hypoglossal Nerve Stimulation Outcomes: A Multicenter Cohort Study. Laryngoscope. 2021 Jul;131(7):1676-1682. doi: 10.1002/lary.29396. Epub 2021 Jan 14. PMID 33443811
- [Background] Nord RS, Fitzpatrick T 4th, Pingree G, Islam A, Chafin A. Should lateral wall collapse be a contraindication for hypoglossal nerve stimulation? Am J Otolaryngol. 2024 Jan-Feb;45(1):104053. doi: 10.1016/j.amjoto.2023.104053. Epub 2023 Sep 24. PMID 37769502
- [Background] Op de Beeck S, Vena D, Mann D, et al. Identifying the site and pattern of pharyngeal collapse using polysomnographic airflow shapes. Sleep Medicine. 2022/12/01/ 2022;100:S252-S253. doi:https://doi.org/10.1016/j.sleep.2022.05.681
- [Background] Op De Beeck S, Vena D, Mann D, et al. Polysomnographic Airflow Shapes and Site of Collapse During Drug-Induced Sleep Endoscopy. C98 DEEP PHENOTYPING FOR SLEEP APNEA THERAPY SUCCESS. American Thoracic Society; 2022:A4817-A4817. American Thoracic Society International Conference Abstracts.
- [Background] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467
- [Background] Safiruddin F, Vanderveken OM, de Vries N, Maurer JT, Lee K, Ni Q, Strohl KP. Effect of upper-airway stimulation for obstructive sleep apnoea on airway dimensions. Eur Respir J. 2015 Jan;45(1):129-38. doi: 10.1183/09031936.00059414. Epub 2014 Sep 3. PMID 25186270
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Lou B, Rusk S, Nygate YN, Quintero L, Ishikawa O, Shikowitz M, Greenberg H. Association of hypoglossal nerve stimulator response with machine learning identified negative effort dependence patterns. Sleep Breath. 2023 May;27(2):519-525. doi: 10.1007/s11325-022-02641-y. Epub 2022 May 27. PMID 35622197

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT06372847/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT06372847/ICF_001.pdf